CLINICAL TRIAL: NCT05495841
Title: OPTiMASK: Comparison of Pre-oxygenation With Standard Face Mask Combined With High Flow Nasal Oxygen With Pre-oxygenation With Standard Face Mask Alone
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Talmor, Anesthesia Department Chair, Beth Israel Deaconess Medical Center
Other Study IDs: 2022P000396
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Face Mask Alone: 40 patients receiving the pre-oxygenation face mask alone method during clinical routine will be studied. As per clinical standard, the standard oxygen facemask will be tightly applied on the face of the patient at 100% FiO2 for 3 to 4 minutes. In case of suspected full stomach, it is recommended to perform a rapid sequence induction and the patient does not receive bag-mask ventilation during the apnea period (45-60s). In the other case, a standard pre-oxygenation will be performed (see figure 1: experimental design of the study).
  Interventions: Device: Pre-oxygenation
- Face Mask and Nasal Cannula: 40 patients using the pre-oxygenation combined facemask + HFNO technique as part of routine clinical care will be studied. As to clinical standards, the standard oxygen facemask will be tightly applied on the face of the patient at 100% FiO2 for 3 to 4 minutes and HFNO at 100% with a flow at 40 L/minutes during the pre-oxygenation (the flow can be decreased to less than 40 L/minutes if no tolerance by the patient). Then, after a general anesthesia induction and/or a rapid sequence induction is performed, the patient receives HFNO at 100% FiO2 and the flow of HFNO is increased to up to 80 L/minutes (which corresponds to a close delivered FiO2 at 80%) during the apnea period (1 to 2 min) until correct position of the endotracheal tube is confirmed with capnography.
  Interventions: Device: Pre-oxygenation

INTERVENTIONS:
Device: Pre-oxygenation — Process of administrating oxygen prior to intubation

SUMMARY:
This is an observational, prospective study of patients undergoing a surgical procedure. Three parallel studies are taking place with collaborators in other countries. This study aims to bring novel insights regarding the benefits of pre-oxygenation combining standard oxygen facemask with high-flow nasal oxygen (HFNO), as opposed to standard oxygen facemask alone by assessing end-tidal oxygen (ETO2) levels after intubation.

DETAILED DESCRIPTION:
This is an observational, prospective study of patients undergoing a surgical procedure. A total of 80 patients will be enrolled at BIDMC. Patients meeting inclusion criteria with no exclusions will be approached for consent. 40 patients receiving the pre-oxygenation face mask alone method during clinical routine and 40 patients using the pre-oxygenation combined facemask + HFNO technique as part of routine clinical care will be studied. No randomization will be employed. Choice of pre-oxygenation approach is at the discretion of the clinician. Patients will be enrolled as a convenience sample, such that the first 40 patients will be those with face mask alone, and the second 40 will be patients with face mask + HFNO. Research assistants will discuss the pre-oxygenation plan with the anesthesiologist as part of the screening process. Data will be collected including EtO2 levels during two minutes following intubation.

Methodology

1. Face mask alone: As per clinical standard, the standard oxygen facemask will be tightly applied on the face of the patient at 100% FiO2 for 3 to 4 minutes. In case of suspected full stomach, it is recommended to perform a rapid sequence induction and the patient does not receive bag-mask ventilation during the apnea period (45-60s). In the other case, a standard pre-oxygenation will be performed (see figure 1: experimental design of the study).
2. Face mask + Nasal cannula: As to clinical standards, the standard oxygen facemask will be tightly applied on the face of the patient at 100% FiO2 for 3 to 4 minutes and HFNO at 100% with a flow at 40 L/minutes during the pre-oxygenation (the flow can be decreased to less than 40 L/minutes if no tolerance by the patient). Then, after a general anesthesia induction and/or a rapid sequence induction is performed, the patient receives HFNO at 100% FiO2 and the flow of HFNO is increased to up to 80 L/minutes (which corresponds to a close delivered FiO2 at 80%) during the apnea period (1 to 2 min) until correct position of the endotracheal tube is confirmed with capnography.

Assessments The study does not require any research procedures other than passive data collection. For this study, EtO2 levels will be recorded at more frequent intervals than what is entered in the anesthesia record. Therefore, study staff will collect these data from the anesthesia machine in the operating room, where values are displayed on a breath-by-breath basis

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* All consecutive patients for scheduled or non-scheduled surgery with or without indication of rapid sequence induction (full-stomach)
* Undergoing general anesthesia with orotracheal intubation

Exclusion Criteria:

* Age < 18 years
* Hemodynamic instability
* Intubation without laryngoscopy (i.e., fiberoptic intubation for anticipated "cannot ventilate situation" or mouth opening < 2 cm), facial surgery
* Adults subject to legal protection
* Pregnancy (due to higher risk of oxygen desaturation and aspiration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study accepts patients undergoing a surgical procedure. Patients would be considered for eligibility regardless of race, ethnicity or gender.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Lowest EtO2 value | start of intubation to 2 minutes after
  Lowest EtO2 value within the two minutes following tracheal intubation

SECONDARY OUTCOMES:
SpO2 at the start and at the end of the procedure | start of intubation to 4 minutes after
  SpO2 at the start and at the end of the procedure and EtO2 each minute during the four minutes of pre-oxygenation
Tolerance of the device | entirety of procedure
  Tolerance of the device (discomfort considered if the patient asks for reduction of the gas flow of HFNC: Yes or No
Lowest SpO2 | start of intubation to 2 minutes after
  Lowest SpO2 during intubation and within 2 min after intubation
Highest level of EtCO2 | start of intubation to 2 minutes after
  Highest level of EtCO2 within 2 min following intubation
Rate of oxygen desaturation | entirety of procedure
  Rate of oxygen desaturation below 95% during the procedure
Number of laryngoscopy attempts | before surgical procedure
  Number of laryngoscopy attempts before successful tracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Talmor, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This study will conduct anonymous data collection in order to ensure the anonymity of each person participating in the study. No information allowing the identification of persons will be communicated to third parties.

REFERENCES:
- [Derived] Jaber S, De Jong A, Schaefer MS, Zhang J, Ma X, Hao X, Zhou S, Lv S, Banner-Goodspeed V, Niu X, Sfara T, Talmor D. Preoxygenation with standard facemask combining apnoeic oxygenation using high flow nasal cannula versuss standard facemask alone in patients with and without obesity: the OPTIMASK international study. Ann Intensive Care. 2023 Apr 4;13(1):26. doi: 10.1186/s13613-023-01124-x. PMID 37014462